CLINICAL TRIAL: NCT03949660
Title: Targeting Improvements in Bowel Function and Quality of Life Using Epidural Stimulation and Training After Severe Spinal Cord Injury
Brief Title: Improving Bowel Function and Quality of Life After Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Charles Hubscher, Assistant Professor, University of Louisville
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 19.0435
Record Dates: First submitted 2019-05-07; First posted 2019-05-14 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Neurogenic Bowel
Keywords: bowel; spinal cord injury; epidural stimulation
MeSH Terms: conditions — Neurogenic Bowel; Spinal Cord Injuries | interventions — Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Epidural stimulation for blood pressure without stand (Experimental): To assess whether epidural stimulation, used for regulating blood pressure without standing, is neuromodulatory for bowel motility after motor complete SCI
  Interventions: Device: Stimulation for blood pressure without stand
- Epidural stimulation for blood pressure with stand (Experimental): To assess whether epidural stimulation, used for regulating blood pressure with standing, is neuromodulatory for bowel motility after motor complete SCI
  Interventions: Device: Stimulation for blood pressure with stand
- Epidural stimulation for trunk and core without stand (Experimental): To assess whether epidural stimulation, used for activating the trunk and core musculature without standing, is neuromodulatory for bowel evacuation after motor complete SCI
  Interventions: Device: Stimulation for trunk and core without stand
- Epidural stimulation for trunk and core with stand (Experimental): To assess whether epidural stimulation, used for activating the trunk and core musculature with standing, is neuromodulatory for bowel evacuation after motor complete SCI
  Interventions: Device: Stimulation for trunk or core with stand

INTERVENTIONS:
Device: Stimulation for blood pressure without stand — Consists of 80 daily training sessions using epidural stimulation optimized for blood pressure for up to 6 hours of stimulation a day.
  Arms: Epidural stimulation for blood pressure without stand
Device: Stimulation for blood pressure with stand — Consists of 80 daily sessions similar to the 1st intervention (without stand) plus 2 hours of epidural stimulation optimized for stand training.
  Arms: Epidural stimulation for blood pressure with stand
Device: Stimulation for trunk and core without stand — Consists of 80 daily training sessions using epidural stimulation optimized for trunk/core/voluntary function for up to 6 hours of stimulation a day.
  Arms: Epidural stimulation for trunk and core without stand
Device: Stimulation for trunk or core with stand — Consists of 80 daily sessions similar to the 1st intervention (without stand) plus 2 hours of epidural stimulation optimized for stand training.
  Arms: Epidural stimulation for trunk and core with stand

SUMMARY:
Bowel dysfunction is consistently rated as one of the most common complications affecting daily life for individuals with spinal cord injury. The overall objective of this study is to investigate whether the use of specific spinal cord epidural stimulation will affect bowel function. This study will also examine how alterations in bowel function influence quality of life outcomes. The results of this study may aid in the development of treatments to help individuals with spinal cord injuries that have impaired bowel function.

DETAILED DESCRIPTION:
Participants in this study must be enrolled in the TS - EPI study (IRB# 16.0179) which provides the spinal cord epidural implant and training interventions. You will receive two sets of interventions, each one lasting 80 sessions for a total of 160 sessions. Assessments for bowel function and quality of life will be performed as part of this study and are conducted at baseline/pre-training, post-Intervention 1, post-Intervention 2, and at the 6-month and 12-month follow-ups. Your participation in this study will last up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at the time of enrollment
* At least 2 years post injury
* Non-progressive spinal cord injury
* Stable medical condition
* Unable to voluntarily move all joints of the legs
* Unable to stand independently
* Cardiovascular dysfunction including presence of persistent resting low blood pressures and/or symptoms of autonomic dysreflexia and/or orthostatic hypotension and/or dysregulation in response to postural changes and/or highly variable blood pressures in 24 hour period
* Bowel dysfunction as a result of spinal cord injury

Exclusion Criteria:

* Ventilator dependent
* Untreated painful musculoskeletal dysfunction, unhealed fracture or pressure sore
* Untreated psychiatric disorder or ongoing drug abuse
* Colostomy bag
* Any implanted pump (i.e., baclofen pump, pain pump, etc)
* Cardiovascular or bowel dysfunction unrelated to SCI
* Ongoing nicotine use
* Pregnant at the time of enrollment or planning to become pregnant during the time course of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-09-15 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Wireless Motility Capsule | Change from Baseline after 4 months, 8 months, 14 months, 20 months.
  Use of the FDA approved SmartPill and device to record information about motility.
Ambulatory blood pressure and heart rate monitoring | Change from Baseline after 4 months, 8 months, 14 months, 20 months.
  Blood pressure will be recorded over a 24-hour period of time outside the lab using a flexible finger cuff on your non-dominant hand.
Anorectal Manometry (ARM) | Change from Baseline after 4 months, 8 months, 14 months, 20 months.
  While lying on your side, while a small, flexible tube, about the size of a thermometer, with a balloon at the end will be inserted into the rectum.
  The catheter is connected to equipment that measures pressure. A small balloon attached to the catheter may be inflated in the rectum to assess muscle responses.
  You will be asked to relax, squeeze, and push at various times. The anal sphincter muscle pressures are measured during each of these muscle contraction/relaxation actions.
  Surface patch EMG electrodes will be placed near the buttocks to evaluate muscle activity of the anal sphincter.
Bowel Diary | Change from Baseline after 4 months, 8 months, 14 months, 20 months.
  Keep a log of various aspects of your bowel program, including how often and how long it takes you to complete your program.
International spinal cord injury bowel function basic data set (Version 2.0) | Change from Baseline after 4 months, 8 months, 14 months, 20 months.
  Complete a short questionnaire about your bowel management. 16 items: date of data collection, gastrointestinal and anal sphincter dysfunction unrelated to SCI, surgical procedures on the gastrointestinal tract, defecation method and bowel-care procedures, average time required for defecation, frequency of defecation, uneasiness, headache or perspiration during defecation, digital stimulation or evacuation of the anorectum, frequency of fecal incontinence, flatus incontinence, need to wear pad or plug, oral laxatives and prokinetics, anti-diarrheal agents, perianal problems, abdominal pain and discomfort and the neurogenic bowel dysfunction score are computed by adding the points given in parenthesis after each relevant variable in the data-set. Total score range is from (0-45). Total neurogenic bowel score (optional): 0-6 Very minor, 7-9 Minor, 10-13 Moderate, 14 or more, Severe neurogenic bowel dysfunction.
Quality of Life Questionnaire measured with the Spinal Cord Injury - Quality of Life (SCI-QOL) items relevant to bowel management. | Change from Baseline after 4 months, 8 months, 14 months, 20 months.
  Complete a series of short questionnaires about your quality of life. SCI-QOL measurements scores range from (0-100). It includes 19 calibrated items banks and 3 fixed length scales spanning the broad domains of physical-medical health, emotional health, social participation and physical functioning.
Interviews | Change from Baseline after 4 months, 8 months, 14 months, 20 months.
  Interviews about your perspective on changes in bowel management and recovery throughout the study, conducted by a qualitative researcher.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Frazier Rehab Institute, Louisville, Kentucky
  - University of Louisville, Louisville, Kentucky

IPD SHARING:
Plan to Share IPD: No